CLINICAL TRIAL: NCT01283425
Title: An Open-label, Randomized, Two-period Crossover Study to Evaluate the Safety Use of the InsuPatch Device in Daily Life Conditions.
Brief Title: Evaluation of the Safety Use of the InsuPatch Device in Daily Life Conditions
Acronym: Daily Life
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insuline Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G080106/B
Record Dates: First submitted 2011-01-19; First posted 2011-01-26 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: MiniMed Paradigm insulin pump; insulin Lispro; Insulin Aspart; Quick-set infusion set
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): InsuPatch use for 3 months.
  Interventions: Device: InsuPatch
- Control (No Intervention)

INTERVENTIONS:
Device: InsuPatch — Heaters for single use and a permanent control unit.
  Arms: Test

SUMMARY:
The study is an open-label, randomized, two-period crossover study. Up to one hundred and twenty (120) subjects with type 1 diabetes mellitus (T1DM) who use the MiniMed paradigm insulin pump, who meet the inclusion/exclusion criteria and who provide written Informed Consent will be enrolled in the study. The aim of the study is to examine the safety of the InsuPatch device in a home use setting. Mild Hypoglycemia,hyperglycemia and Adverse events will be compared between two phases of the study : 3 months with the use of the device and 3 months without the use of the device.

DETAILED DESCRIPTION:
The primary objective of this study is to show that safety parameters are similar, when delivering insulin subcutaneously in subjects with type I diabetes using the InsuPatch device along with the Medtronic Minimed Paradigm insulin infusion pump and the Medtronic Minimed Quick-Set® infusion set compared to subcutaneous insulin delivered with the above mentioned equipment, without the InsuPatch device.

The participation of each subject in this study will be up to seven months and will include three phases: one week Run in phase , 3 months with device use and 3 months without device use. Study will include 4 clinic visits and bi weekly calls. During the entire study the subjects will be requested to preform at least 5 blood glucose self measurements and record results in a logbook.At each visit blood will be drawn for HBA1C test.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age range 18- 65 years old (including 18 and 65 years old)
2. BMI: 18-35 kg/m2
3. Type 1 diabetes patients using a MiniMed Paradigm insulin pump for at least six months, who are administering insulin Lispro or Insulin Aspart and are using the Quick-set infusion set.
4. Patients with T1DM whose HbA1c values are at or below 9.5% (including 9.5%) and at or above 6% (including 6%).
5. Agree to sign consent form before any study-specific tests or procedures are to be performed.
6. Subject's completed at least 14 measurements during the Run-In Phase and readiness to continue the study with at least 5 blood glucose recordings per day and keep a logbook during the study period.
7. Subject readiness to use the InsuPatch, his comprehension of the study requirements and treatment procedures.
8. Willingness to comply with all specified follow-up evaluations.

Exclusion Criteria:

1. Pregnancy
2. Breast feeding women.
3. Alcohol addiction
4. CABG (Coronary Artery Bypass Graft), MI (Myocardial Infarction) or active Ischemic Heart Disease prior to study date.
5. CVA (cardiovascular accident) or TIA (transient ischemic accident) events prior to study date.
6. Uncontrolled hypertension (blood pressure in mm HG >160 systolic or > 95 diastolic) .
7. Any history of gastroparesis or enteroparesis.
8. Abnormal kidney and/ or liver function tests. (Defined as Creatinine >1.5 mg/dL, liver tests> 2 times the upper limit of normal).
9. A severe hypoglycemic event requiring a glucagon injection or intravenous glucose infusion within the last six months prior to study inclusion.
10. Hypoglycemia unawareness.
11. Diabetic ketoacidosis (severe, with hospitalization) within the last six months prior to study inclusion.
12. Psychological incompetence.
13. Signs of drug abuse.
14. Any other clinical condition or history, which seems to be relevant for the Principle Investigator to disqualify a participant.
15. Subjects with diminished skin integrity, Excessive fibrosis, lipo-hypertrophy or eczema at infusion sites.
16. Heat sensitive subjects.
17. Subjects involved in or planning to participate in other studies.
18. Subjects using any drug therapy, other than insulin, to control their blood glucose levels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
frequency of mild hypoglycemia events (Blood Glucose<60mg/dl) with InsuPatch and without. | safety will be assesed after 6 months at the study completion
  The confirmatory safety endpoint is, for each subject, frequency of mild hypoglycemia events (Blood Glucose<60mg/dl) with InsuPatch and without.
  The number of events will be assessed from subject logbook and will be compared between two arms.

SECONDARY OUTCOMES:
Frequency of hyperglycemic events (BG>300 mg/dl, Fasting BG>250 mg/dl) with InsuPatch and without. | safety will be assesed after 6 months at the study completion
  Frequency of hyperglycemic events (BG>300 mg/dl, Fasting BG>250 mg/dl) with InsuPatch and without.The number of events will be assesed from subject logbook and will be compared between two arms.
Adverse events (AE's) count with InsuPatch and without. | safety will be assesed after 6 months at the study completion
  Adverse events (AE's) whether or not deemed related to study device with InsuPatch and without.The number of events will be assesed dering the subject visits and bi-weekly calls and will be compared between two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Wainstein Julio, MD, Principal Investigator — Wolfsom Medical Center, Holon, Israel; Itamar Raz, MD, Principal Investigator — Hadassah Medical Organization; Klonoff David, MD, Principal Investigator — Mills Peninsula Health Services; Naim Shhada, MD, Principal Investigator — Rambam Health Care Campus; Orit Hamiel, MD, Principal Investigator — Sheba Medical Center; Moshe Philips, MD, Principal Investigator — Schnieder Children's Medical Center; Anat Yaffe, Md, Principal Investigator — Hiullel Yaffe Medical Center
Locations (8):
- Mills-Peninsula Health Services, San Mateo, California, United States
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe, Hadera
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Haddasah Medical Organization, Jerusalem
  - Schneider Children's hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan

REFERENCES:
- See also: Related Info — http://www.insuline-medical.com